CLINICAL TRIAL: NCT05447650
Title: Microcurrent Stimulation Therapy for Nonexudative Age-related Macular Degeneration (i-SIGHT): A Multicenter, Randomized, Sham-controlled, Feasibility Device Trial.
Brief Title: Microcurrent Stimulation Therapy for Nonexudative Age-related Macular Degeneration (i-SIGHT)
Acronym: i-SIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i-Lumen Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ILS-AMD-201
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Age-Related Macular Degeneration; Dry Age-related Macular Degeneration; Nonexudative Age-related Macular Degeneration
Keywords: AMD; Dry AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- i-Lumen AMD Active (Experimental): Active transpalpebral microcurrent stimulation therapy
  Interventions: Device: i-Lumen(TM) AMD
- i-Lumen AMD Sham (Sham Comparator): Sham transpalpebral microcurrent stimulation therapy
  Interventions: Device: i-Lumen(TM) AMD Sham

INTERVENTIONS:
Device: i-Lumen(TM) AMD — Transpalpebral microcrurrent stimulation
  Arms: i-Lumen AMD Active
Device: i-Lumen(TM) AMD Sham — Transpalpebral sham stimulation
  Arms: i-Lumen AMD Sham

SUMMARY:
Evaluate the safety and efficacy of transpalpebral microcurrent stimulation (MCS) therapy for patients with nonexudative (dry) age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
The i-Lumen(TM) AMD device is for in-office therapy use to deliver microcurrent electrical stimulation transpalpebrally (via the eyelid) for use by an ophthalmologist. The i-Lumen AMD device contains proprietary software with preset treatment algorithms and is calibrated at each session to the individual participant.

Up to 30 enrolled participants will be randomized (2:1 active to sham ratio) and complete the initial 5-day loading treatment sessions. Participants completing the initial loading sessions will receive two (2) days of maintenance treatments and be following and be followed through the one (1) year time point.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥50 years.
* Non-exudative age-related macular degeneration defined as AREDS category 3 Intermediate AMD and/or geographic atrophy
* Best-corrected distance visual acuity 20/40 to 20/200 (inclusive) in the study eye, and BCVA 20/100 or better in the fellow eye

Key Exclusion Criteria:

* History and/or evidence of exudative age-related macular degeneration in either eye
* History and/or evidence of diabetic retinopathy in either eye
* Current tobacco or tobacco-related product use or history within the past 10 years of heavy smoking (on average, more than half a pack of cigarettes per day)
* Central chorioretinal atrophy in the study eye
* Glaucoma in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Adverse Device Effects | Through study completion, Month 12 timepoint
  Incidence of device- and/or treatment-related serious adverse events (SAEs) and/or serious adverse device effects (SADE) at any point during the study

OTHER OUTCOMES:
Mean change best corrected distance visual acuity | Through Month 12 timepoint
  Mean change from baseline of best corrected distance visual acuity (CDVA) letter score

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Mundy, Study Director — i-Lumen Scientific, Inc.
Locations (10):
- United States (10):
  - Associated Retina Consultants, Phoenix, Arizona
  - Bay Area Retina Associates, Walnut Creek, California
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Cumberland Valley Retina Consultants, Chambersburg, Pennsylvania
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Charles Retina Institute, Germantown, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Star Retina, Burleson, Texas
  - Texas Retina Associates, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No